CLINICAL TRIAL: NCT01460810
Title: A Prospective Pilot Study of Surgical Radiation Shielding With Vitrectomy & Silicone Oil Tamponade for the Protection of Radiation-induced Ocular Injury in the Treatment of Choroidal Melanoma With Radioactive Iodine-125 Plaque Brachytherapy
Brief Title: Safety and Efficacy of Silicone Oil Tamponade for Surgical Attenuation of Radiation Damage in Choroidal Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11-0366
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Choroidal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1000CsK Silicon Oil Tamponade (Experimental): In 20 patients, a standard three-port vitrectomy will be performed. Following a standard air-fluid exchange, the eye will be filled with Silikon-1000 silicone oil in standard fashion. At a subsequent surgery, a standard two-port pars plana vitrectomy will be performed to remove the silicone oil and replace it with saline. The removed silicone oil will be tested onsite for traces of radiation.
  Interventions: Other: 1000CsK Silicon Oil Tamponade

INTERVENTIONS:
Other: 1000CsK Silicon Oil Tamponade — Details covered in arm description

SUMMARY:
A prospective, experimental, case series of 20 patients, with choroidal melanoma, in which pars plana vitrectomy and Silicone oil as vitreous substitute will be used as intraocular shielding for attenuating the deleterious effects of radiation dose delivered to healthy ocular tissue during Iodine-125 plaque brachytherapy treatment and assess if the treatment can reduce the incidence and severity of radiation-induced adverse effects like radiation retinopathy and permanent loss of vision.

DETAILED DESCRIPTION:
Melanoma arising from the choroid and ciliary body is the most common primary intraocular cancer. The Collaborative Ocular Melanoma Study (COMS) randomized clinical trial of I-125 brachytherapy versus enucleation for medium-sized choroidal melanoma (2.5-10.0 mm in thickness and ≤ 16 mm in diameter) showed that, for patients who met the eligibility criteria, there was no statistically significant difference in all-cause mortality between I-125 brachytherapy and enucleation 5, 10, and 12 years following treatment. The COMS trial supported the use of globe-conserving I-125 brachytherapy. Following brachytherapy, however, visual acuity in the treated eye generally declined at a rate of approximately 2 lines of visual acuity per year and nearly 45% of patients lost ambulatory vision (≤20/200) in the treated eye by 3 years.

Adverse effects of plaque brachytherapy include cataract, radiation-associated proliferative retinopathy, maculopathy and papillopathy. Radiation maculopathy, which may result in decreased central vision, cystoid macular edema (CME), macular ischemia, and chorioretinal atrophy, was reported in other series in 18% to 43% of treated eyes within 5 years after brachytherapy. Typical onset occurred 18-24 months following treatment. Primary risk factors for radiation papillopathy and maculopathy were total radiation dose to the affected structures, proximity of the tumor to the affected structures and systemic conditions such as diabetes mellitus. No treatment for radiation maculopathy or papillopathy has been proven to be effective in a randomized clinical trial.

Radiation injury to vital structures may be avoided or shielded with the use of materials such as lead that have a higher effective atomic number and density than tissue. However, solid metals are not amenable to use within the eye (Figure 1).

There have been previous efforts to try to use a vitreous substitute in order to protect intraocular structures from the deleterious effects of radiations. In an animal study, Finger et al, demonstrated that iodinated contrast agents (iophendylate, iohexol, and iopamidol) could block radiation intraocularly. But these substances were highly toxic and could not be retained in the eye due to high water solubility.

The technique of vitrectomy and oil tamponade during plaque brachytherapy has been performed previously in humans by Dr. Tara McCannel at UCLA. During a paper presentation at the 2010 meeting of the American Society of Retina Specialist in Vancouver, BC, the first series of 10 patients were presented, and no complications of the technique were reported. It is now a commonly applied technique at this center for treatment of choroidal melanoma (Oncology Times 2010; 32(14):36, UCLA, Clinical Update 2011; 20(1):1, 4)

In this prospective pilot study the investigators propose that patients will undergo standard plaque placement for treatment of their ocular melanoma in addition to pars plana vitrectomy and silicone oil infusion. When patients return for their scheduled plaque removal one week later, they will also undergo removal of the silicone oil from the eye. Placement of silicone oil should not alter the radiation dose delivered to the tumor, as there is no physical space between the tumor and the radioactive plaque for silicone oil to be present. The reduction in radiation to healthy ocular structures by using the oil technique may be sufficient to avoid the clinical complications caused by radiation-induced injury.

ELIGIBILITY:
Inclusion Criteria:

* All treatment-naïve patients with clinical diagnosis of primary choroidal melanoma, amenable to treatment with plaque brachytherapy, aged 18 or older regardless gender, race/ethnicity or existing medical condition unless they are specifically mentioned as exclusion criteria.
* Patients with best corrected visual acuity of 20/400 or better in the study eye.
* Patients in whom the calculated dose of radiation to the optic nerve or macula is > 25 Gray (Gy).

Tumor inclusion criteria:

* Unilateral choroidal melanoma, medium size as defined by COMS classification:

  1. At least 2.5 mm in height, but no more than 10 mm in height (no more than 8.0 mm whenever the tumor was near the optic disc), and
  2. No more than 16.0 mm In diameter, regardless the shape by ultrasound.

Exclusion Criteria:

* History of previous treatment for the choroidal melanoma.
* Pregnancy.
* Patients with any impairment which prevent attending follow-up appointments.
* The presence of concomitant significant life-treating medical conditions that significantly reduces the life expectancy to less than three years.
* The presence of other vision-treating ophthalmic condition, not directly related with choroidal melanoma which is likely to going to require intraocular surgery in the next three years.
* Clinical or radiological evidence of the presence of metastatic disease.
* The presence of significant media opacity (e.g. cataract) that precludes the investigator's ability to grade the tumor, performs retina surgery, or performs follow-up assessments.
* Patients that do not accept the informed consent

Tumor exclusion criteria:

* Inability to successfully grade, stage and delineate the tumor by ultrasound.
* Tumor location that will prevent the correct placement of the plaque or have significant risk of optic nerve damage during plaque placement.
* Tumors that involved the anterior chamber angle, the iris or have detectable extrascleral extension.
* Tumor margin location < 1000 µm from the fovea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Vision Loss | 1 year
  The loss of 5 or more letters from the base line on an Early Treatment Diabetic Retinopathy Study (ETDRS) chart after 1 and 2 years of follow-up.

SECONDARY OUTCOMES:
Severe Visual Loss | 3 years
  The loss of 15 or more letters from base line on and ETDRS chart after three years of follow-up. Contrast sensitivity loss: the loss of 2 or more lines on a Pelli-Robson Chart after 1 and 2 years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Oliver, MD, Principal Investigator — University of Colorado, Denver; Raul Velez-Montoya, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Eye Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Data will be released in publications, but no information will be used that could disclose the subjects' identity.

REFERENCES:
- [Background] Melia BM, Abramson DH, Albert DM, Boldt HC, Earle JD, Hanson WF, Montague P, Moy CS, Schachat AP, Simpson ER, Straatsma BR, Vine AK, Weingeist TA; Collaborative Ocular Melanoma Study Group. Collaborative ocular melanoma study (COMS) randomized trial of I-125 brachytherapy for medium choroidal melanoma. I. Visual acuity after 3 years COMS report no. 16. Ophthalmology. 2001 Feb;108(2):348-66. doi: 10.1016/s0161-6420(00)00526-1. PMID 11158813
- [Background] Quivey JM, Char DH, Phillips TL, Weaver KA, Castro JR, Kroll SM. High intensity 125-iodine (125I) plaque treatment of uveal melanoma. Int J Radiat Oncol Biol Phys. 1993 Jul 15;26(4):613-8. doi: 10.1016/0360-3016(93)90277-3. PMID 8330990
- [Background] Oliver SC, Young TA, Kobe LH, Leu MY, Lee SP, Chun MW, Straatsma BR. Assessment of central vision and macular structure in patients undergoing iodine-125 brachytherapy for ciliochoroidal melanoma. Am J Clin Oncol. 2008 Oct;31(5):488-92. doi: 10.1097/COC.0b013e31816d1c94. PMID 18838887
- [Background] Diener-West M, Earle JD, Fine SL, Hawkins BS, Moy CS, Reynolds SM, Schachat AP, Straatsma BR; Collaborative Ocular Melanoma Study Group. The COMS randomized trial of iodine 125 brachytherapy for choroidal melanoma, III: initial mortality findings. COMS Report No. 18. Arch Ophthalmol. 2001 Jul;119(7):969-82. doi: 10.1001/archopht.119.7.969. PMID 11448319
- [Background] Oittinen HA, O'Shaughnessy M, Cullinane AB, Keohane C. Malignant melanoma of the ciliary body presenting as extraocular metastasis in the temporalis muscle. J Clin Pathol. 2007 Jul;60(7):834-5. doi: 10.1136/jcp.2005.033613. Epub 2007 Jun 1. No abstract available. PMID 17545559
- [Background] Collaborative Ocular Melanoma Study Group.. Assessment of metastatic disease status at death in 435 patients with large choroidal melanoma in the Collaborative Ocular Melanoma Study (COMS): COMS report no. 15. Arch Ophthalmol. 2001 May;119(5):670-6. doi: 10.1001/archopht.119.5.670. PMID 11346394
- [Background] Shields JA, Augsburger JJ, Brady LW, Day JL. Cobalt plaque therapy of posterior uveal melanomas. Ophthalmology. 1982 Oct;89(10):1201-7. doi: 10.1016/s0161-6420(82)34658-8. PMID 7155529
- [Background] Augsburger JJ, Gamel JW, Sardi VF, Greenberg RA, Shields JA, Brady LW. Enucleation vs cobalt plaque radiotherapy for malignant melanomas of the choroid and ciliary body. Arch Ophthalmol. 1986 May;104(5):655-61. doi: 10.1001/archopht.1986.01050170045019. PMID 3518677
- [Background] Adams KS, Abramson DH, Ellsworth RM, Haik BG, Bedford M, Packer S, Seddon J, Albert D, Polivogianis L. Cobalt plaque versus enucleation for uveal melanoma: comparison of survival rates. Br J Ophthalmol. 1988 Jul;72(7):494-7. doi: 10.1136/bjo.72.7.494. PMID 3415941
- [Background] Oliver SC, Leu MY, DeMarco JJ, Chow PE, Lee SP, McCannel TA. Attenuation of iodine 125 radiation with vitreous substitutes in the treatment of uveal melanoma. Arch Ophthalmol. 2010 Jul;128(7):888-93. doi: 10.1001/archophthalmol.2010.117. PMID 20625051
- [Background] Finger PT, Ho TK, Fastenberg DM, Hyman RA, Stroh EM, Packer S, Perry HD. Intraocular radiation blocking. Invest Ophthalmol Vis Sci. 1990 Sep;31(9):1724-30. PMID 2211021
- [Background] Soheilian M, Mazareei M, Mohammadpour M, Rahmani B. Comparison of silicon oil removal with various viscosities after complex retinal detachment surgery. BMC Ophthalmol. 2006 May 31;6:21. doi: 10.1186/1471-2415-6-21. PMID 16737520
- [Background] Halberstadt M, Domig D, Kodjikian L, Koerner F, Garweg JG. PVR recurrence and the timing of silicon oil removal. Klin Monbl Augenheilkd. 2006 May;223(5):361-6. doi: 10.1055/s-2006-926594. PMID 16705505
- [Background] Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010 Jul 10;376(9735):124-36. doi: 10.1016/S0140-6736(09)62124-3. Epub 2010 Jun 26. PMID 20580421
- [Background] Rizzo S, Belting C, Genovesi-Ebert F, di Bartolo E. Incidence of retinal detachment after small-incision, sutureless pars plana vitrectomy compared with conventional 20-gauge vitrectomy in macular hole and epiretinal membrane surgery. Retina. 2010 Jul-Aug;30(7):1065-71. doi: 10.1097/IAE.0b013e3181cd48b0. PMID 20616684
- [Background] Jones S, Edwards RT. Diabetic retinopathy screening: a systematic review of the economic evidence. Diabet Med. 2010 Mar;27(3):249-56. doi: 10.1111/j.1464-5491.2009.02870.x. PMID 20536486
- [Background] Polak BC, Crijns H, Casparie AF, Niessen LW. Cost-effectiveness of glycemic control and ophthalmological care in diabetic retinopathy. Health Policy. 2003 Apr;64(1):89-97. doi: 10.1016/s0168-8510(02)00143-4. PMID 12644331
- [Background] Palmer AJ, Weiss C, Sendi PP, Neeser K, Brandt A, Singh G, Wenzel H, Spinas GA. The cost-effectiveness of different management strategies for type I diabetes: a Swiss perspective. Diabetologia. 2000 Jan;43(1):13-26. doi: 10.1007/s001250050003. PMID 10672449